CLINICAL TRIAL: NCT00508469
Title: Adherence of Patients Using Travalert® for Instillation of a Fixed Combination of Travoprost 0.004%/Timolol 0.5% Compared to a Concomitant Regimen of Travoprost 0.004% and Timolol 0.5%
Brief Title: Adherence Assessment With Travalert Dosing Aid
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Alcon Research (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: EMD-06-03
Record Dates: First submitted 2007-07-26; First posted 2007-07-30 (Estimated); Results first posted 2012-07-12 (Estimated); Last update posted 2012-07-12 (Estimated); Status verified 2012-06

CONDITIONS: Open-angle Glaucoma; Ocular Hypertension
Keywords: Intraocular pressure; Open-angle glaucoma; Ocular hypertension; Adherence; Compliance
MeSH Terms: conditions — Glaucoma, Open-Angle; Ocular Hypertension; Patient Compliance | interventions — Travoprost; Timolol; Duotrav; Ophthalmic Solutions

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Travalert with travoprost/timolol fixed combination (Experimental): One drop in the study eye once daily at 9 p.m. for six months using the Travalert device.
  Interventions: Drug: Travoprost 0.004%/timolol 0.5% fixed combination eye drops (DuoTrav); Device: Travalert Dosing Aid
- Travalert with travoprost and timolol (Experimental): One drop travoprost in the study eye at 9 p.m. and one drop of timolol in the study eye twice daily (9 a.m. and 9 p.m.) for six months using a separate Travalert device for each medication.
  Interventions: Drug: Travoprost 0.004% eye drops; Drug: Timolol 0.05% eye drops; Device: Travalert Dosing Aid

INTERVENTIONS:
Drug: Travoprost 0.004%/timolol 0.5% fixed combination eye drops (DuoTrav) — One drop in the study eye once daily at 9 p.m. for six months using the Travalert device.
  Other Names: DuoTrav®
  Arms: Travalert with travoprost/timolol fixed combination
Drug: Travoprost 0.004% eye drops — One drop in the study eye once daily at 9 p.m. for six months using the Travalert device.
  Arms: Travalert with travoprost and timolol
Drug: Timolol 0.05% eye drops — One drop in the study eye twice daily at 9 a.m. and 9 p.m. for six months using the Travalert device.
  Arms: Travalert with travoprost and timolol
Device: Travalert Dosing Aid — Approved device used with study medication to record time of instillation and quantify dosing

SUMMARY:
The purpose of the study is to compare adherence in patients on a fixed combination of travoprost 0.004%/timolol 0.5% and patients on a concomitant combination of travoprost 0.004% and timolol 0.5% using the Travalert® device.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of open-angle glaucoma or ocular hypertension;
* Inadequate control with beta-blocker or prostaglandin monotherapy and starting therapy with travoprost 0.004% and timolol 0.05%;
* Intraocular pressure (IOP) at the screening visit in at least one eye ≥ 19 mmHg but not exceeding 36 mmHg in either eye;
* Other protocol-defined inclusion criteria may apply.

Exclusion Criteria:

* Females of childbearing potential currently pregnant, breastfeeding, or not taking control measures to prevent pregnancy;
* Not currently receiving treatment for lowering IOP with beta-blockers or prostaglandin analogs;
* Currently on therapy or was in therapy with another investigational agent within 30 days prior to the baseline visit;
* History of chronic or recurrent severe inflammatory eye disease, or history of ocular trauma within the past six (6) months, or history of ocular infection or ocular inflammation within the past three (3) months in either eye;
* History of clinically significant or progressive retinal disease or history of any other severe ocular pathology in either eye that would preclude the administration of a topical prostaglandin analogue;
* History of severe or serious hypersensitivity to prostaglandin drugs or their analogues, to topical or systemic beta-blockers, or to any components of the study medication;
* Intraocular surgery within the past six (6) months or ocular laser surgery within the past three (3) months as determined by patient history and/or examination in either eye;
* Any abnormality preventing reliable applanation tonometry of either eye;
* Best-corrected visual acuity worse than 20/30 Snellen in either eye;
* Use of any additional topical or systemic ocular hyposensitive medication during the study;
* Other protocol-defined exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2007-10; Primary Completion 2010-01 (Actual); Study Completion 2010-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Dr Francisco M. Honrubia, Study Director — Independent
Locations (1):
- Zaragoza, Zaragoza, Spain

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from 5 hospitals in Spain.
Pre-assignment Details: Baseline characteristics are presented for the per-protocol population.
Period: Overall Study
Arm/Group | Travalert With Travoprost/Timolol Fixed Combination | Travalert With Travoprost and Timolol
Started | 52 | 50
Completed | 35 | 40
Not Completed | 17 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Travalert With Travoprost/Timolol Fixed Combination | Travalert With Travoprost and Timolol | Total
Number analyzed (Participants) | 43 | 42 | 85
Age Continuous [Mean (Standard Deviation); unit: years] | 63.8 (11.1) | 68.6 (11.8) | 66.2 (11.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 25 | 51
  Male | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Adherence
Description: Patients were considered adherent if a minimum of 80% of their instillations were administered ±2 hours of the scheduled time.
Time Frame: 6 months
Population: Per protocol
Measure: Number; unit: percentage of adherent patients
Arm/Group | Travalert With Travoprost/Timolol Fixed Combination | Travalert With Travoprost and Timolol
Number analyzed (Participants) | 43 | 42
percentage of adherent patients | 63 | 43

ADVERSE EVENTS:
Time Frame: Adverse events were collected for the duration of the study: 2 years, 3 months.
Description: The safety population includes all enrolled patients.
Arm/Group | Travalert With Travoprost/Timolol Fixed Combination | Travalert With Travoprost and Timolol
Serious Adverse Events (participants affected / at risk) | 1/52 | 1/50
Other Adverse Events (participants affected / at risk) | 0/52 | 0/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Travalert With Travoprost/Timolol Fixed Combination (N=52) | Travalert With Travoprost and Timolol (N=50)
Heart Failure (Cardiac disorders) | 1 (1) | 0 (0)
Brachycardia (Cardiac disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other